CLINICAL TRIAL: NCT02123602
Title: The Effects of a Trunk Strengthening Program on Anterior Knee Pain in an Adolescent Athletic Population: a Randomized Clinical Trial
Brief Title: Core Stabilization for the Treatment of Anterior Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Kenneth Learman, Associate Professor of Physical Therapy, Youngstown State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #093-2014
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; abdominal muscles
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Core stabilization (Experimental): This arm will receive 3 weeks of core stabilization training followed by 3 weeks of lower extremity stretching and strengthening as appropriate to address impairments noted in the examination and to progress function.
  Interventions: Other: core stabilization
- Lower extremity training only (Active Comparator): This arm with receive 6 weeks of impairment based stretching and strengthening to restore function.
  Interventions: Other: lower extremity training only

INTERVENTIONS:
Other: core stabilization
  Arms: Core stabilization
Other: lower extremity training only
  Arms: Lower extremity training only

SUMMARY:
The investigators hypothesize that the use of trunk (core) stabilization exercises early in treatment combined with lower extremity exercises will enhance the outcome over lower extremity exercises alone in the treatment of young athletes with anterior knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 13-20 years of age clinically diagnosed with anterior knee pain.
* Pain should be peripatellar and should include at least 3 of the following:

  1. experienced during or after activity
  2. prolonged sitting
  3. with stair climbing or descending
  4. squatting
  5. kneeling.
* The subject should be active for at least 30 minutes per day.

Exclusion Criteria:

* Previous knee surgery
* Signs and symptoms of a specific structural diagnosis not consistent with AKP such as meniscal, ACL, PCL, or collateral ligament tears, pain referral from hip or lumbar spine (determined during examination), traumatic patellar dislocation, an inability to adequately understand or communicate in English.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-07 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Lower extremity functional scale | 6 weeks
  LEFS is a functional scale that estimates how much the subject's function is disrupted by their condition.

SECONDARY OUTCOMES:
Kujala anterior knee pain scale | 6 weeks
  The Kujala scale measures the amount and impact of anterior knee pain on the subject's life
Patient specific functional scale | 6 weeks
  The PSFS rates subject's ability to do the 3 functional activities that are bothered the most by the knee pain
Numeric pain rating scale | 6 weeks
  The NPRS measures the subject's current knee pain

OTHER OUTCOMES:
Global rating of change | 6 weeks
  The GRoC measures the subject's overall estimation of improvement.
Self-reported percent recovery | 6 weeks
  The subject reports their estimated overall percentage of improvement from the start of care

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Learman, PhD, PT, Principal Investigator — Youngstown State University
Locations (1):
- Poland Medical Center, Poland, Ohio, United States

REFERENCES:
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] van Linschoten R, van Middelkoop M, Berger MY, Heintjes EM, Verhaar JA, Willemsen SP, Koes BW, Bierma-Zeinstra SM. Supervised exercise therapy versus usual care for patellofemoral pain syndrome: an open label randomised controlled trial. BMJ. 2009 Oct 20;339:b4074. doi: 10.1136/bmj.b4074. PMID 19843565
- [Background] Collins NJ, Bisset LM, Crossley KM, Vicenzino B. Efficacy of nonsurgical interventions for anterior knee pain: systematic review and meta-analysis of randomized trials. Sports Med. 2012 Jan 1;42(1):31-49. doi: 10.2165/11594460-000000000-00000. PMID 22149696
- [Background] Earl JE, Hoch AZ. A proximal strengthening program improves pain, function, and biomechanics in women with patellofemoral pain syndrome. Am J Sports Med. 2011 Jan;39(1):154-63. doi: 10.1177/0363546510379967. Epub 2010 Oct 7. PMID 20929936
- [Background] Koumantakis GA, Watson PJ, Oldham JA. Trunk muscle stabilization training plus general exercise versus general exercise only: randomized controlled trial of patients with recurrent low back pain. Phys Ther. 2005 Mar;85(3):209-25. PMID 15733046